CLINICAL TRIAL: NCT01500720
Title: Randomized Phase II Study of Cabazitaxel Versus Topotecan in Small Cell Lung Cancer Patients With Progressive Disease During or After a First Line Platinum Based Chemotherapy
Brief Title: Cabazitaxel Compared to Topotecan for the Treatment of Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARD12166; 2011-003415-31 (EudraCT Number); U1111-1123-3503 (Other: UTN)
Record Dates: First submitted 2011-12-22; First posted 2011-12-28 (Estimated); Results first posted 2015-04-13 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-03

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — cabazitaxel; XRP6258; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cabazitaxel (Experimental)
  Interventions: Drug: Cabazitaxel
- Topotecan (Active Comparator)
  Interventions: Drug: Topotecan

INTERVENTIONS:
Drug: Cabazitaxel — Cabazitaxel 25 milligram per square meter (mg/m^2) intravenously (IV) on Day 1 every 3 weeks (21-day cycle) until unacceptable toxicity, disease progression or withdrawal consent.
  Other Names: XRP6258
  Arms: Cabazitaxel
Drug: Topotecan — Topotecan 1.5 mg/m^2 IV on Day 1 to Day 5 every 3 weeks (21-Day cycle) until unacceptable toxicity, disease progression or withdrawal consent.
  Arms: Topotecan

SUMMARY:
Primary Objective:

To demonstrate progression free survival (PFS) improvement for cabazitaxel compared to topotecan in participants with sensitive or resistant/refractory small cell lung cancer following a first line platinum based chemotherapy.

Secondary Objectives:

* To assess disease progression free rate at 12 weeks
* To assess Response Rate (Response Evaluation Criteria in Solid Tumor [RECIST] 1.1) and duration of response
* To assess Overall Survival (OS)
* To assess the Safety (National Cancer Institute - Common Toxicity Criteria [NCI-CTC] version 4.03)
* To assess the Health-Related Quality of Life (HRQoL)

DETAILED DESCRIPTION:
Participants are to be treated until progressive disease, unacceptable toxicity or refusal for further study treatment.

All participants are to be followed for disease progression documentation and for participant status until the study cut-off date.

ELIGIBILITY:
Inclusion criteria :

* Histological/cytological proven locally advanced or metastatic small cell lung cancer with progressive disease during or after first line platinum based chemotherapy
* Male or female greater than or equal to (>=) 18 years (or country's legal age of majority if greater than [>]18 years)
* Participants with measurable disease, Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.1)
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to (<=) 1

Exclusion criteria:

* Absence of signed and dated Institutional Review Board (IRB)-approved participant informed consent form prior to enrollment into the study
* More than one prior chemotherapy regimen. Prior treatment with topotecan or taxanes
* Less than 28 days elapsed from prior treatment with chemotherapy, radiotherapy or surgery to the time of randomization (Radiotherapy for bone pain palliation is allowed)
* Adverse events (excluding alopecia) from any prior anticancer therapy of grade >1 (National Cancer Institute Common Terminology Criteria [NCI CTCAE] v4.03) at the time of randomization
* Uncontrolled Central Nervous System (CNS) metastases: participants with CNS metastases may have previous irradiation, only participants with stable disease or response to irradiation who are without CNS symptoms and on a maximum steroid dose of dexamethasone 8 mg daily or equivalent could be included
* Participants with known leptomeningeal metastases
* History of other, invasive neoplasm requiring ongoing therapy
* Participation in another clinical trial and any concurrent treatment with any investigational drug within 30 days prior to randomization
* Any of the following within 6 months prior to study enrollment: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, New York Heart Association class III or IV congestive heart failure, stroke or transient ischemic attack
* Any severe acute or chronic medical condition, which could impair the ability of the participant to participate in the study or interfere with interpretation of study results
* Known Human Immunodeficiency Virus (HIV) disease, or active hepatitis B or C (systematic testing was not required)
* Pregnant or breast-feeding woman. Positive serum or urine pregnancy test prior to randomization
* Participant with reproductive potential (M/F) who did not agree to use an accepted and effective method of contraception during the study treatment period and for at least 6 months after the completion of the study treatment. The definition of "effective method of contraception" was based on the investigator's judgment. Effective method of contraception should also be adapted to local regulation
* History of hypersensitivity to polysorbate 80
* Inadequate organ and bone marrow function as evidenced by:

  * Hemoglobin less than [<] 9.0 gram per deciliter (g/dL)
  * Absolute neutrophil count <1.5 x 10^9 per liter
  * Platelet count <100 x 10^9 per liter
  * Aspartate Aminotransferase/Serum Glutamic Oxaloacetic Transaminase (AST/SGOT) and/or alanine aminotransferase/Serum Glutamic-Pyruvic Transaminase (ALT/SGPT) >2.5 x Upper Limit of Normal (ULN)
  * Alkaline Phosphatase (AP) >2.5 x ULN. In case of liver metastases AP >5 x ULN
  * Total bilirubin >1.0 x ULN
  * Serum Creatinine >1.5 x ULN. If creatinine 1.0 - 1.5 x ULN, creatinine clearance will be calculated according to Chronic Kidney Disease Epidemiology Collaboration formula, and creatinine clearance <60 milliliter per minute (mL/min) was exclude the participant.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2012-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (58):
- United States (5):
  - Investigational Site Number 840007, Muscle Shoals, Alabama
  - Investigational Site Number 840005, Omaha, Nebraska
  - Investigational Site Number 840006, Lebanon, New Hampshire
  - Investigational Site Number 840003, Middletown, Ohio
  - Investigational Site Number 840001, Philadelphia, Pennsylvania
- Investigational Site Number 076001, Porto Alegre, Brazil
- Canada (4):
  - Investigational Site Number 124003, Montreal
  - Investigational Site Number 124002, Oshawa
  - Investigational Site Number 124004, Rimouski
  - Investigational Site Number 124001, Toronto
- Chile (2):
  - Investigational Site Number 152001, Santiago
  - Investigational Site Number 152005, Santiago
- France (6):
  - Investigational Site Number 250005, Brest
  - Investigational Site Number 250004, Caen
  - Investigational Site Number 250006, La Tronche
  - Investigational Site Number 250002, Lille
  - Investigational Site Number 250003, Saint-Herblain
  - Investigational Site Number 250007, Villejuif
- Germany (2):
  - Investigational Site Number 276003, Großhansdorf
  - Investigational Site Number 276006, Löwenstein
- Greece (5):
  - Investigational Site Number 300005, Athens
  - Investigational Site Number 300003, Athens
  - Investigational Site Number 300001, Heraklion
  - Investigational Site Number 300002, Thessaloniki
  - Investigational Site Number 300004, Thessaloniki
- Hungary (4):
  - Investigational Site Number 348001, Budapest
  - Investigational Site Number 348004, Budapest
  - Investigational Site Number 348002, Budapest
  - Investigational Site Number 348003, Törökbálint
- Italy (4):
  - Investigational Site Number 380001, Genova
  - Investigational Site Number 380002, Livorno
  - Investigational Site Number 380005, Novara
  - Investigational Site Number 380004, Parma
- Norway (3):
  - Investigational Site Number 578001, Oslo
  - Investigational Site Number 578003, Stavanger
  - Investigational Site Number 578002, Trondheim
- Poland (4):
  - Investigational Site Number 616004, Gdansk
  - Investigational Site Number 616003, Lublin
  - Investigational Site Number 616002, Poznan
  - Investigational Site Number 616001, Warsaw
- Romania (4):
  - Investigational Site Number 642003, Cluj-Napoca
  - Investigational Site Number 642005, Cluj-Napoca
  - Investigational Site Number 642001, Craiova
  - Investigational Site Number 642002, Timișoara
- Russia (4):
  - Investigational Site Number 643001, Moscow
  - Investigational Site Number 643005, Saint Petersburg
  - Investigational Site Number 643006, Tula
  - Investigational Site Number 643003, Yaroslavl
- South Korea (3):
  - Investigational Site Number 410001, Seoul
  - Investigational Site Number 410003, Seoul
  - Investigational Site Number 410002, Seoul
- Spain (4):
  - Investigational Site Number 724002, Badalona
  - Investigational Site Number 724004, Barcelona
  - Investigational Site Number 724005, Málaga
  - Investigational Site Number 724001, Valencia
- Ukraine (3):
  - Investigational Site Number 804002, Dnipropetrovsk
  - Investigational Site Number 804004, Donetsk
  - Investigational Site Number 804001, Lviv

REFERENCES:
- [Derived] Beaumont H, Evans TL, Klifa C, Guermazi A, Hong SR, Chadjaa M, Monostori Z. Discrepancies of assessments in a RECIST 1.1 phase II clinical trial - association between adjudication rate and variability in images and tumors selection. Cancer Imaging. 2018 Dec 11;18(1):50. doi: 10.1186/s40644-018-0186-0. PMID 30537991
- [Derived] Evans TL, Cho BC, Udud K, Fischer JR, Shepherd FA, Martinez P, Ramlau R, Syrigos KN, Shen L, Chadjaa M, Wolf M. Cabazitaxel Versus Topotecan in Patients with Small-Cell Lung Cancer with Progressive Disease During or After First-Line Platinum-Based Chemotherapy. J Thorac Oncol. 2015 Aug;10(8):1221-8. doi: 10.1097/JTO.0000000000000588. PMID 26200278

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 232 participants were screened of which 53 were screen failure and 179 were randomized.
Groups:
- Cabazitaxel: Cabazitaxel (XRP6258) 25 milligram per square meter (mg/m^2) intravenously (IV) on Day 1 every 3 weeks (21-day cycle) until unacceptable toxicity, disease progression or withdrawal consent.
Period: Overall Study
Arm/Group | Cabazitaxel | Topotecan
Started | 90 (Randomized) | 89 (Randomized)
Treated | 89 | 88
Completed | 85 (Cancer progression,adverse event,consent withdrawal are considered as completed(defined in protocol)) | 80 (Cancer progression,adverse event,consent withdrawal are considered as completed(defined in protocol))
Not Completed | 5 | 9
Not completed — Randomized But Not Treated | 1 | 1
Not completed — Other | 4 | 8

BASELINE CHARACTERISTICS:
Population: Randomized population included all randomized participants, and was analyzed according to the randomized treatment.
Groups:
- Cabazitaxel: Cabazitaxel 25 mg/m^2 IV on Day 1 every 3 weeks (21-day cycle) until unacceptable toxicity, disease progression or withdrawal consent.
- Total: Total of all reporting groups
Arm/Group | Cabazitaxel | Topotecan | Total
Number analyzed (Participants) | 90 | 89 | 179
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (9.4) | 61.6 (10.0) | 60.7 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 27 | 54
  Male | 63 | 62 | 125
Race/Ethnicity, Customized [Number; unit: participants]
  Race: Caucasian/White | 80 | 82 | 162
  Race: Black | 1 | 2 | 3
  Race: Asian/Oriental | 9 | 4 | 13
  Race: Other | 0 | 1 | 1
  Ethnicity: Hispanic | 4 | 3 | 7
  Ethnicity: Not Hispanic | 86 | 86 | 172
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — ECOG criteria:
  * 0: Fully active
  * 1: Ambulatory, carry out work of a light or sedentary nature
  * 2: Ambulatory, capable of all selfcare
  * 3: Capable of limited selfcare, confined to bed or chair more than 50% of waking hours
  * 4: Completely disabled, no selfcare, totally confined to bed or chair
  * 5: Dead
  participants
    0 | 31 | 17 | 48
    1 | 59 | 71 | 130
    2 | 0 | 1 | 1
Primary Tumor Site [Number; unit: participants]
  Lungs | 16 | 20 | 36
  Right Lung | 33 | 43 | 76
  Left Lung | 40 | 26 | 66
  Other: Mediastino-Hilar | 1 | 0 | 1
Stage at Diagnosis [Number; unit: participants] — Disease stages were decided based on tumor size, lymph nodes and metastasis (as per National Comprehensive Cancer Network guidelines Version 2.2013).
  participants
    IIA | 1 | 1 | 2
    IIB | 2 | 1 | 3
    IIIA | 2 | 12 | 14
    IIIB | 25 | 15 | 40
    IV | 57 | 55 | 112
    Unknown | 3 | 5 | 8
Number of Organs Involved [Mean (Standard Deviation); unit: organs] | 3.6 (1.3) | 3.8 (1.4) | 3.7 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time interval from the date of randomization to the date of occurrence of the first documented tumor progression or death due to any cause, whichever came first. Median PFS was estimated using the Kaplan-Meier method. Progression was defined using Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.1) as: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study or unequivocal progression of existing non-target lesion. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeter (mm). The appearance of one or more new lesions is also considered progression.
Time Frame: Randomization to first tumor progression/clinical deterioration or death (maximum 7.6 months)
Population: Intent-to-treat (ITT) population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabazitaxel | Topotecan
Number analyzed (Participants) | 90 | 89
months | 1.4 [1.4 to 1.5] | 3.0 [2.7 to 4.1]
Statistical Analysis 1: Comparison: Cabazitaxel vs Topotecan; Test type: Superiority or Other; p < 0.0001, Stratified Two-Sided Log-Rank Test — P-value was calculated from stratified two-sided log-rank test, stratifying for brain metastases and lactate dehydrogenase (LDH) level at the time of randomization; Cox Proportional Hazard = 2.169, 95% CI 2-sided [1.563 to 3.01] — Hazard ratio was estimated using a COX Proportional Hazards regression model, stratifying for brain metastases and LDH level at the time of randomization

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time interval from the date of randomization to the date of death due to any cause. In the absence of confirmation of death, survival time was to be censored at the last date the participant was known to be alive. Median time was estimated by Kaplan-Meier curve.
Time Frame: From randomization to date of death (maximum 15 months)
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabazitaxel | Topotecan
Number analyzed (Participants) | 90 | 89
months | 5.2 [3.38 to 6.11] | 6.8 [5.03 to 8.08]

3. Secondary Outcome: Progression Free Rate at Week 12
Description: Progression was defined using Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.1) as: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study or unequivocal progression of existing non-target lesion. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression. Death due to disease progression within 12 weeks without radiological documentation of progressive disease was counted as an event. Percentage of participants who were progression free at week 12 are reported.
Time Frame: Week 12
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cabazitaxel | Topotecan
Number analyzed (Participants) | 90 | 89
percentage of participants | 18.9 [11.4 to 28.5] | 52.8 [41.9 to 63.5]

4. Secondary Outcome: Overall Objective Tumor Response Rate
Description: Overall objective tumor response was defined as the proportion of participants with confirmed RECIST 1.1 achieving a complete response (CR) or partial response (PR). CR was defined as disappearance of all target/non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Percentage of participants with overall objective tumor response is reported.
Time Frame: Randomization to disease progression/occurrence (maximum 7.6 months)
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cabazitaxel | Topotecan
Number analyzed (Participants) | 90 | 89
percentage of participants | 0 [0.0 to 4.9] | 10.1 [4.5 to 19.0]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form until 30 days after last study treatment administration (maximum 66 weeks) regardless of seriousness or relationship to investigational product.
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'on treatment period' (from the first study treatment administration until 30 days after the last dose of study treatment). Safety population all randomized participants who received at least one dose of study medication (treated).
Arm/Group | Cabazitaxel | Topotecan
Serious Adverse Events (participants affected / at risk) | 36/89 | 41/88
Other Adverse Events (participants affected / at risk) | 67/89 | 75/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cabazitaxel (N=89) | Topotecan (N=88)
Neutropenic infection (Infections and infestations) | 4 | 5
Neutropenic sepsis (Infections and infestations) | 3 | 1
Bronchitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 6
Postoperative wound infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 10
Neutropenia (Blood and lymphatic system disorders) | 2 | 2
Anaemia (Blood and lymphatic system disorders) | 1 | 6
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 10
Pancytopenia (Blood and lymphatic system disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Paraparesis (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 2 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 2
Hypotension (Vascular disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary microemboli (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Disease progression (General disorders) | 6 | 4
Asthenia (General disorders) | 2 | 2
Death (General disorders) | 1 | 0
Generalised oedema (General disorders) | 1 | 0
Performance status decreased (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 2
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cabazitaxel (N=89) | Topotecan (N=88)
Anaemia (Blood and lymphatic system disorders) | 4 | 18
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 6
Leukopenia (Blood and lymphatic system disorders) | 1 | 6
Neutropenia (Blood and lymphatic system disorders) | 2 | 20
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 14
Decreased appetite (Metabolism and nutrition disorders) | 16 | 13
Dizziness (Nervous system disorders) | 2 | 5
Headache (Nervous system disorders) | 6 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 21
Abdominal pain (Gastrointestinal disorders) | 9 | 3
Abdominal pain upper (Gastrointestinal disorders) | 5 | 2
Constipation (Gastrointestinal disorders) | 8 | 9
Diarrhoea (Gastrointestinal disorders) | 18 | 9
Nausea (Gastrointestinal disorders) | 14 | 11
Stomatitis (Gastrointestinal disorders) | 8 | 3
Vomiting (Gastrointestinal disorders) | 15 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 6
Asthenia (General disorders) | 10 | 17
Fatigue (General disorders) | 26 | 22
Non-cardiac chest pain (General disorders) | 6 | 6
Oedema peripheral (General disorders) | 1 | 5
Pyrexia (General disorders) | 4 | 7
Neutrophil count decreased (Investigations) | 3 | 6
Weight decreased (Investigations) | 7 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.